CLINICAL TRIAL: NCT01860196
Title: A Placebo Controlled, Cross-over, Double Blind, Randomized, Clinical Trial to Compare the Efficacy and Safety of Meditoxin® Injection for Cervical Dystonia in Adults With Cerebral Palsy
Brief Title: Efficacy and Safety of Meditoxin® Injection for Cervical Dystonia in Adults With Cerebral Palsy
Acronym: ATHETOID_CD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Keewon Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT_IT_009
Record Dates: First submitted 2013-05-13; First posted 2013-05-22 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Adult Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment-Placebo Group (Active Comparator): Treatment on 0 day Placebo at 5th week
  Interventions: Drug: Meditoxin
- Placebo-Treatment Group (Active Comparator): Placebo on 0 day Treatment at 5th week
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Meditoxin
  Arms: Treatment-Placebo Group
Drug: Normal saline
  Arms: Placebo-Treatment Group

SUMMARY:
This study aimed to compare the efficacy and safety of Meditoxin® injection for cervical dystonia in adults with cerebral palsy. It is a placebo controlled, Cross-over, Double blind, Randomized, Clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult cerebral palsy patients over 20 years old
* Clinically diagnosed for cervical dystonia more than a year ago
* No improvement with antispasmodics for the last month
* Actively participated and gave informed consent

Exclusion Criteria:

* Allergic to the botulinum toxin
* Limited range of motion in cervical spine
* Patients with fever, infection, cancer, uncontrollable seizure
* Generalized neuromuscular junction disease patients
* Pregnant or breast feeding women, or anticipating pregnancy until 12 weeks after the study stopped
* Patients enrolled in other studies
* History of dose change in 4 weeks: antispasmodics, benzodiazepine, anticholinergics
* Botulinum toxin injection history in 6 months
* Previous history of intrathecal baclofen, selective peripheral denervation, deep brain stimulation
* Otherwise clinically non-eligible patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | 0, 16, 32 weeks
  Change of Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) from baseline TWSTRS at 0 week.

SECONDARY OUTCOMES:
Pain in numerical rating scale (NRS) | Every 4 weeks, up to 32 weeks
  Pain in numerical rating scale (NRS)
Japanese Orthopaedic Association (JOA) score | Every 4 weeks, up to 32 weeks
  Change of Japanese Orthopaedic Association (JOA) score from baseline Japanese Orthopaedic Association (JOA) score at 0 week.
Goal attainment scale | 4, 12, 20, 28 weeks
  Goal attainment scale of subjective improvement from the baseline status at 0 and 16 weeks.

OTHER OUTCOMES:
Adverse effect | Every 4 weeks, up to 32 weeks
  vital sign, adverse effect
computed tomography (CT) | 0, 32 weeks
  Change of cervical spine computed tomography (CT) from baseline CT at 0 week.
videofluoroscopic swallowing study (VFSS) | 0, 12, 28 weeks
  Change of videofluoroscopic swallowing study (VFSS) from baseline VFSS at 0 week.
Blood/Urine laboratory tests | 0, 16, 32 weeks
  1. Hemoglobin, Hematocrit, RBC, WBC, WBC different cell count, Platelet
  2. Alkaline phosphatase, BUN, Creatinine, SGPT(ALT), SGOT(AST), Albumin, Total protein, Total bilirubin, Uric acid, Glucose, Cholesterol, LDH, Na, Ca, K, Cl
  3. Urine pH, Protein, Glucose, Bilirubin, Blood, WBC